CLINICAL TRIAL: NCT03405766
Title: Barriers in the Process of Achieving Informed Consent From Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Akershus (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Sigrid Beitland, Principal investigator, Oslo University Hospital
Other Study IDs: REK 2017/1254
Record Dates: First submitted 2017-12-13; First posted 2018-01-23 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Critically Ill; Ethics; Informed Consent; Study Recruitment
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will explore barriers in the process of achieving informed consent from critically ill patients

DETAILED DESCRIPTION:
The barriers will be divided into four major categories:

* Practical barriers
* Medical barriers
* Legal barriers
* Ethical barriers

ELIGIBILITY:
Inclusion Criteria:

* Patients considered for inclusion in the NORIDES study

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care unit patients
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Study recruitment barriers, Medical | 2018-2022
  Number (%) of patients unable to give consent or to sign
Study recruitment barriers, Ethical | 2018-2022
  Number (%) of patients not asked to give consent due to ethical issues

SECONDARY OUTCOMES:
Study recruitment barriers, Practical | 2018-2022
  Number (%) of cases where practical reasons made consent impossible
Study recruitment barriers, Legal | 2018-2022
  Number (%) of patients where legal issues made consent impossible

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Not planned to share data

REFERENCES:
- [Derived] Dahlberg J, Eriksen C, Robertsen A, Beitland S. Barriers and challenges in the process of including critically ill patients in clinical studies. Scand J Trauma Resusc Emerg Med. 2020 Jun 8;28(1):51. doi: 10.1186/s13049-020-00732-x. PMID 32513204